CLINICAL TRIAL: NCT01903590
Title: PROSPECTIVE RANDOMIZED STUDY COMPARING TVT AND TOT IN FEMALE STRESS URINARY INCONTINENCE WITH NO INTRINSIC SPHINCTER DEFICIENCY
Brief Title: TVT Versus TOT in Urinary Stress Incontinence With No Intrinsic Sphincter Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Sabri Cavkaytar, Obstetrics and Gynecology specialist, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZTB-070713; ZekaiTahirBurak-SCavkaytar1 (Registry Identifier: ZekaiTahirBurak)
Record Dates: First submitted 2013-07-13; First posted 2013-07-19 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-03

CONDITIONS: Female Urinary Stress Incontinence
Keywords: TVT,TOT,Randomized

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transvaginal Tape Surgery (Active Comparator): Randomized 50 patients undergoing TVT
  Interventions: Procedure: TVT surgery TOT surgery
- Transobturator tape surgery (Experimental): Randomized 50 patients undergoing TOT
  Interventions: Procedure: TVT surgery TOT surgery

INTERVENTIONS:
Procedure: TVT surgery TOT surgery

SUMMARY:
The aim of this study is to compare trans-vaginal tape(TVT) and trans-obturator tape(TOT) procedure in female urinary stress incontinence with no intrinsic sphincter deficiency.

DETAILED DESCRIPTION:
Patients with isolated stress incontinence attending to Dr Zekai Tahir Burak Woman Health Teaching and Research Hospital Urogynecology Department will be prospectively randomized,by a computer generated randomisation code,to the TVT or TOT. The patients will be aware of the type of the surgical procedure before the operation.

Preoperative evaluation includes clinical history,urinanalysis,pelvic examination QoL assessment and urodynamic study. QoL included Urogenital Distress Inventory Short Form (UDI-6) and the Incontinence Impact Questionnaire Short Form( IIQ-7).Urodynamic study includes cystometry,urethral profilometry and Valsalva leak point pressure (VLPP).In all patients,pelvic floor defect will be evaluated according to the POP quantification (POPQ) staging.To diagnose the occult stress incontinence in patients with pelvic prolapse, a cough test after reducing the prolapse will be performed.Patients will be followed up at 6 and 12 months postoperatively.Objective cure is defined as a negative cough stress test .Negative cough stress test ,but occasional urine leakage during stress will be considered ''improved''.

Postoperative subjective outcomes will be categorized as follows:cured (UDI-6 and IIQ-7 postoperative<10), improved (UDI-6 and IIQ-7 if postoperative>preoperative) and worsened (UDI-6 and IIQ-7 if postoperative<preoperative).

ELIGIBILITY:
Inclusion Criteria:

* Women with urinary stress incontinence with no intrinsic sphincter deficiency
* Women with or without pelvic organ prolapse

Exclusion Criteria:

* Previous incontinence surgery
* Urge incontinence or overactive bladder
* Mixed incontinence
* Intrinsic sphincter deficiency
* Body mass index>35
* Un-willing for randomisation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficiency of TVT and TOT in stress incontinence with no intrinsic deficiency | One year
  Postoperative UDI-6 and IIQ-7 <10 and negative cough test will be defined as ''cured''

SECONDARY OUTCOMES:
Objective effectiveness by cough test at 6 and 12 th months postoperatively | One year
  A patient with a bladder filled 300 cc saline will cough and if no leakage of urine,the patient will be described as ''cured''.
Subjective effectiveness by UDI-6 and IIQ-7 at 6-12 th months postoperatively | One year
  Postoperative subjective outcomes will be categorized as follows:cured (UDI-6 and IIQ-7 postoperative<10), improved (UDI-6 and IIQ-7 if postoperative>preoperative) and worsened (UDI-6 and IIQ-7 if postoperative<preoperative).
Short term and long term surgical complications | One year
  Bleeding,bladder and bowel perforation,mesh erosion etc..
The prevalence of voiding dysfunction at 1 and 12 th months postoperatively | One year
  Postoperative residual volume after first voiding >100 cc ,difficulty in voiding will be described as ''voiding dysfunction''.

CONTACTS AND LOCATIONS:
Overall Officials: Sabri Cavkaytar, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Dr Zekai Tahir Burak Woman Health Teaching and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)